CLINICAL TRIAL: NCT05504356
Title: Volunteers to Investigate Best Results for Ablation and Novel Therapies for Atrial Fibrillation
Acronym: VIBRANT-AF
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: American College of Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: P0548846
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
VIBRANT-AF seeks to:

* Identify clinically relevant predictors of effectiveness and complications of AF ablation procedures in a prospective, US-based, multi-center, real-world longitudinal study
* Assess changes in modifiable lifestyle-related exposures influence the effectiveness of AF ablation
* Determine incidence and predictors of complications of AF ablation procedures

Participants will connect with the Eureka Research Platform and answer a series of surveys and activities over a one-year period. They will be asked about lifestyle habits, recurrence of AFib, hospitalizations, and general feelings and emotions.

DETAILED DESCRIPTION:
Catheter ablation for Atrial Fibrillation is the most commonly performed cardiac electrophysiology procedure. Although now standard of care in professional society guidelines, recommendations favoring the procedure are predominately based on randomized trials or single-center experiences from high-volume institutions staffed by expert operators. Participants enrolled in those randomized trials are healthier than those undergoing the procedure in the "real world," and the actual experiences of patients throughout the US are not represented by those referred to tertiary-referral centers that most frequently publish their retrospective observations. Although administrative databases provide a glimpse into what happens in the real-world, ICD-9, ICD-10, and CPT codes cannot capture specific procedural approaches or patient perspectives. For this reason, this study aims to leverage the Eureka Research Platform, a digital health infrastructure to enable longitudinal follow-up and ascertainment of patient reported outcomes.

This is a longitudinal, observational cohort study. 15,000 subjects are planned to be enrolled, and will be followed for a period of one year. Subjects will be asked weekly survey questions on weekly habits, complications, medication usage, and hospitalizations. They will have the option to receive AliveCor Kardia devices for remote ECG monitoring, as well as connect their Apple HealthKit data. Surveys will be conducted via the Eureka mobile app.

In conjunction with the Eureka Research Platform, the study will leverage the AF Ablation National Cardiovascular Data Registry (NCDR) run by the American College of Cardiology (ACC). This rapidly growing registry includes comprehensive data regarding patient, procedure, and institution-level characteristics, now includes over 200 institutions around the US, and has already enrolled more than 47,000 patients. However, the registry is limited to data collected during the index procedure visit, without longitudinal follow-up or patient reported outcomes. The study will link the Eureka Research Platform data to NCDR registry data on the index procedure for a subset of participants, allowing for analysis of longitudinal follow-up together with index procedure data.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and older
* Must have a smartphone device (iOS and/or Android) and cell phone number to participate on the mobile app, and will be willing to download the Eureka Research Platform mobile application
* Must have email address to participate on the web portal (accessible on any web-connected device)
* Undergone a catheter ablation procedure for atrial fibrillation in the week prior to recruitment, or have an ablation planned for within a week from recruitment

Exclusion Criteria:

* Unable to consent for themselves
* Unable to read, speak, comprehend English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of AF (i.e. new onset AF, paroxysmal AF, persistent AF, Permanent AF), who have recently or will imminently be undergoing AF ablation. Subjects will be at least 18 years of age or older, and be English-speakers, as well as adhere to the inclusion criteria pertaining to access to the Eureka mobile app (owning a smartphone device and cell phone number, email address)
Sampling Method: Non-Probability Sample
Enrollment: 1125 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to Atrial Fibrillation Recurrence | 1 year
  Time to atrial fibrillation, after employing a 3-month blanking period. Atrial Fibrillation Recurrence includes patient-reported symptoms of AF or Kardia-based ECG evidence of AF.

SECONDARY OUTCOMES:
Mean Change in the Atrial Fibrillation Effect on Quality-of-Life (AFEQT) Score | 6 months, 1 year
  Atrial Fibrillation Effect on Quality-of-Life will be measured using the AFEQT, the score ranges from 0 to 100, with higher scores indicating better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Marcus, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No